CLINICAL TRIAL: NCT06232330
Title: Effects of Task Oriented Approach Versus Rhythmic Initiation And Stabilization Techniques of PNF on Trunk Control in Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of TOA Versus PNF Techniques on Trunk Control in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0738
Record Dates: First submitted 2023-12-26; First posted 2024-01-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: CP; Hemiplegia; Rhythmic Initiation; Rhythmic Stabilization; TOA
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: The study will be randomized clinical trial used to evaluate the effect of task-oriented training on balance in spastic hemiplegic cerebral palsied children. Subjects with hemiplegic Cerebral Palsy meeting the inclusion and exclusion criteria will be divided into two groups using non-probability sampling techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): TOA and conventional therapy
  Interventions: Device: Group A
- Group B (Experimental): PNF and conventional therapy
  Interventions: Device: Group B

INTERVENTIONS:
Device: Group A — This group will receive TOA which include Weight transfers from a standing position and stepping in various star-type directions, Sit-ups from different heights with the hemiplegic lower limb behind the normal lower limb, From a kneeling position alternately projecting the lower limb forward, From a standing position with a limited base of support turning head and trunk right to left, Continuous walking on a treadmill for 10 minutes, Ascending and descending of stairs, Crossing 4 obstacles with continuous walking, Walking while simultaneously pushing a stroller, Walking while holding an object, Walking on different surfaces and slopes, The intervention took place for 5 days a week for 6 week for 20 minutes. Pre measurement was taken before the intervention and after 6 weeks post measurement was taken.
  Arms: Group A
Device: Group B — This group will receive PNF techniques for trunk control. Rhythmic initiation and Rhythmic stabilization for a span of 20 minutes on both sides. In rhythmic initiation patient will move passively from trunk flexion into extension and then back to the flexed position When the patient is relaxed and moving easily, ask for active assisted motion Then begin resisting the motion then patient will perform independently in rhythmic stabilization Resist an isometric contraction of the patient's trunk flexor muscles patient will match the resistance in front and then in back
  Arms: Group B

SUMMARY:
Cerebral palsy occurs in 2-2.5 per 1000 live births, seems to be the most common cause of lifelong physical disability, and has an impact on the child, caregivers, and society. The incidence of cerebral palsy continues to rise owing to the large numbers of premature and high-risk infants who survive. Task-oriented arm approaches promote intensive, meaningful, and goal-oriented training in subjects, and the voluntary functional activities of these subjects possibly reduce their motor disabilities.

DETAILED DESCRIPTION:
The study will be randomized clinical trial used to evaluate the effectiveness of TOA and PNF on trunk control in children with hemiplegic cerebral palsy. Subjects with hemiplegic cerebral palsy meeting the inclusion and exclusion criteria will be divided into two groups using non- probability sampling techniques. Assessment will be done using trunk control measuring scale and pediatric reach test . Group A will receive TOA and conventional therapy and Group B will receive PNF and conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* The level of gross motor function between I and III in accordance with the Gross Motor Function Classification System (GMFCS)
* The degree of spasticity in the affected lower extremity between grade 1 and 1+ in accordance with the Modified Ashworth scale
* 6-12 years of age
* Ability to understand and follow verbal instructions

Exclusion Criteria:

* Surgical procedures within the past 6 months
* Botox injection within 6 months
* Unstable Seizures
* Other comorbidity condition (Multiple Disabilities)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measuring Scale | 6 weeks
  The TCMS scale assesses seated trunk control in three dimensions. The maximum score is 58 points where 20 points correspond to static balance, 28 to selective movement control, and 10 to the ability to perform dynamic reaching. The items are scored from 0 to 3, with 0 being the inability to perform the task and 3 being the complete performance of the item.
Pediatric Reach Test | 6 weeks
  It is used to measure the standing balance in normally developed or children with cerebral palsy, that's why is done in standing position. The standing position will be described first and target will be set under the supervision first forward reach will be tested and after this lateral reach will be tested. Reliability of this test is within rater (0.54, 0.88 ICC) and among the rater is (0.50, 0.93ICC)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Ijaz, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salphale VG, Kovela RK, Qureshi MI, Harjpal P. Effectiveness of Pelvic Proprioceptive Neuromuscular Facilitation on Balance and Gait Parameters in Children With Spastic Diplegia. Cureus. 2022 Oct 22;14(10):e30571. doi: 10.7759/cureus.30571. eCollection 2022 Oct. PMID 36415346